CLINICAL TRIAL: NCT03655301
Title: An Open-label, Non-randomized, Phase I Study to Evaluate the Effect of Copanlisib (a Single Intravenous Dose of 60 mg) on the Pharmacokinetics (PK) and Pharmacodynamics (PD) of Metformin (MATE2-K Substrate) in Healthy Volunteers
Brief Title: Effect of Copanlisib on Metformin Pharmacokinetics and Pharmacodynamics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19951
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Results first posted 2019-12-23 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — copanlisib; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Copanlisib (Aliqopa, BAY80-6946) (Experimental): All subjects will receive a single dose of metformin 1000 mg on Days 1 and 8 in a fasting state. Subjects will also receive a single i.v. dose of 60 mg copanlisib on Day 8 as part of the combination with metformin.
  Interventions: Drug: Copanlisib (Aliqopa, BAY80-6946); Drug: Metformin

INTERVENTIONS:
Drug: Copanlisib (Aliqopa, BAY80-6946) — The copanlisib dose for this study is the standard dose recently approved and also used in Phase 1, 2 and 3 studies across the copanlisib development program: 60 mg i.v. infusion administered intermittently on Days 1, 8 and 15 of a 28-day cycle.
  In this study subjects will receive a single i.v. dose of 60 mg copanlisib on day 8.
Drug: Metformin — Single dose of 1000 mg is administered orally.

SUMMARY:
The purpose of this study is to learn about a drug-drug interaction. When two medications are taken together at the same time, one medication may change the activity of the other medication in the body - this is called a drug-drug interaction. This study is looking at the effect the Bayer study drug, copanlisib, has on metformin, a commonly used medication to treat diabetes. During the study, blood and urine samples will be collected and analyzed to learn about pharmacokinetics (how copanlisib changes metformin levels in the body) and pharmacodynamics (the effect metformin has on the body when taken together with copanlisib) when someone takes both copanlisib and metformin together.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects - as determined by the investigator or medically qualified designee based on medical evaluations, including medical history, physical examination, laboratory tests and cardiac monitoring
* Aged 18 to 45 years at the first screening visit
* Body Mass Index (BMI) of 18.0 - 34 kg / m*2 , with body weight ≥ 50 kg
* Creatinine clearance ≥ 90 mL/min using the Modification of Diet in Renal Disease
* Adequate end organ and bone marrow function

Exclusion Criteria:

* Existing relevant diseases of vital organs (e.g. liver diseases, heart diseases), central nervous system (for example seizures) or other organs (e.g. diabetes mellitus)
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Relevant respiratory insufficiency / disorder
* Administration of strong CYP3A4 inhibitors or inducers within 2 weeks prior to dosing
* Known history of hypersensitivity (or known allergic reaction) to copanlisib, metformin, related compounds, or any components of the formulation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2019-02-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaceutical Product Development (PPD), LLC, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one study center in the US, between 11-Sep-2018 (first participant first visit) and 12-Nov-2018 (last participant last visit).
Pre-assignment Details: A total of 50 participants signed the informed consent form, of them 37 participants were screen failures. The remaining 13 participants received the study treatment.
Groups:
- Copanlisib (Aliqopa, BAY80-6946) + Metformin: Participants received 2 oral doses of metformin, 1 dose (1000 milligram [mg]) on Day 1 and 1 dose (1000 mg) on Day 8, and a single dose of copanlisib (60 mg, 1 h infusion) on Day 8. A wash-out period of 7 days was maintained between the 2 doses of metformin.
Period: Overall Study
Arm/Group | Copanlisib (Aliqopa, BAY80-6946) + Metformin
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safey Analysis Set (SAF): included all participants who received at least one dose of the study medication
Arm/Group | Copanlisib (Aliqopa, BAY80-6946) + Metformin
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: SAF
  Years | 28.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: SAF
  Participants
    Female | 6
    Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: SAF
  Participants
    Hispanic or Latino | 8
    Not Hispanic or Latino | 5
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: SAF
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 6
    White | 7
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Drug Concentration of Metformin in Plasma After Single Dose Administration (Cmax)
Description: Maximum observed drug concentration of metformin in plasma after single dose administration without copanlisib (Day 1) and in combination with copanlisib (Day 8) were measured.
Time Frame: Pre-dose and up to 24 hours after drug administration on Day 1 and Day 8
Population: Pharmacokinetic Analysis Set (PKS): included all participants with a valid PK profile for metformin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Arm/Group | Copanlisib (Aliqopa, BAY80-6946) + Metformin
Number analyzed (Participants) | 13
microgram per liter (mcg/L)
  Day 1 | 1550 (16.4)
  Day 8 | 1460 (27.6)
Statistical Analysis 1: Comparison: Copanlisib (Aliqopa, BAY80-6946) + Metformin; Day 8 (with copanlisib) to Day 1 (without copanlisib) ratio of Cmax; Test type: Other; Least squares mean = 0.9405, 90% CI 2-sided [0.8093 to 1.0931]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to 24 Hours of Metformin After Single Dose Administration (AUC[0-24])
Description: Area under the concentration versus time curve from zero to 24 hours of metformin after single dose administration without copanlisib (Day 1) and in combination with copanlisib (Day 8) were measured.
Time Frame: Pre-dose and up to 24 hours after drug administration on Day 1 and Day 8
Population: Pharmacokinetic Analysis Set (PKS): included all participants with a valid PK profile for metformin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per liter (mcg*h/L)
Arm/Group | Copanlisib (Aliqopa, BAY80-6946) + Metformin
Number analyzed (Participants) | 13
microgram*hour per liter (mcg*h/L)
  Day 1 | 7710 (17.6)
  Day 8 | 8640 (20.8)
Statistical Analysis 1: Comparison: Copanlisib (Aliqopa, BAY80-6946) + Metformin; Day 8 (with copanlisib) to Day 1 (without copanlisib) ratio of AUC(0-24); Test type: Other; Least squares mean = 1.1205, 90% CI 2-sided [1.0000 to 1.2555]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity of Metformin After Single Dose Administration (AUC)
Description: Area under the concentration verus time curve from zero to infinity of metformin after single dose without copanlisib (Day 1) and in combination with copanlisib (Day 8) were measured.
Time Frame: Pre-dose and extrapolated up to infinity after drug administration on Day 1 and Day 8
Population: Pharmacokinetic Analysis Set (PKS) with valid data for this evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per liter (mcg*h/L)
Arm/Group | Copanlisib (Aliqopa, BAY80-6946) + Metformin
Number analyzed (Participants) | 12
microgram*hour per liter (mcg*h/L)
  Day 1 | 8000 (16.9)
  Day 8 | 8900 (21.2)
Statistical Analysis 1: Comparison: Copanlisib (Aliqopa, BAY80-6946) + Metformin; Day 8 (with copanlisib) to Day 1 (without copanlisib) ratio of AUC; Test type: Other; Least squares mean = 1.1147, 90% CI 2-sided [0.9772 to 1.2714]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. Treatment-emergent adverse events (TEAEs) were defined as adverse events that started or worsened after the start of study drug administration up to 30 days after last administration of the study medication.
Time Frame: From start of study medication until 30 days after end of treatment with study medication.
Population: Safety Analysis Set (SAF): included all participants who received at least one dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Copanlisib (Aliqopa, BAY80-6946) + Metformin
Number analyzed (Participants) | 13
Participants
  Day 1 | 5
  Day 8 | 9
  Total | 11

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events by Severity
Description: An adverse event (AE) was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. Treatment-emergent adverse events (TEAEs) were defined as adverse events that started or worsened after the start of study drug administration up to 30 days after last administration of the study medication. TEAEs per severity were reported.
Time Frame: From start of study medication until 30 days after end of treatment with study medication.
Population: Safety Analysis Set (SAF): included all participants who received at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Copanlisib (Aliqopa, BAY80-6946) + Metformin
Number analyzed (Participants) | 13
Participants
  Day 1: Mild | 5
  Day 1: Moderate | 0
  Day 1: No AEs | 8
  Day 8: Mild | 7
  Day 8: Moderate | 2
  Day 8: No AEs | 4
  Total: Mild | 9
  Total: Moderate | 2
  Total: No AEs | 2

6. Secondary Outcome: Plasma Lactate Levels
Description: Lactate levels were analyzed in plasma samples collected during metformin alone or in combination with copanlisib. Plasma lactate levels were summarized by treatment conditions (Day 1 and Day 8).
Time Frame: Up to 24 hours after study drug administration on Day 1 and Day 8
Population: Safety Analysis Set (SAF): included all participants who received at least one dose of the study medication.
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Copanlisib (Aliqopa, BAY80-6946) + Metformin
Number analyzed (Participants) | 13
mmol/L
  Day 1 (0h) | 0.78 [0.5 to 1.1]
  Day 1 (0.5h) | 0.74 [0.4 to 1.0]
  Day 1 (1h) | 0.83 [0.5 to 1.6]
  Day 1 (2h) | 0.74 [0.5 to 1.0]
  Day 1 (4h) | 1.01 [0.6 to 1.7]
  Day 1 (6h) | 0.75 [0.6 to 1.0]
  Day 1 (8h) | 0.80 [0.6 to 1.1]
  Day 1 (12h) | 1.04 [0.7 to 2.4]
  Day 1 (24h) | 0.89 [0.5 to 1.8]
  Day 8 (0h) | 0.78 [0.6 to 1.2]
  Day 8 (0.5h) | 0.85 [0.5 to 1.4]
  Day 8 (1h) | 0.90 [0.6 to 1.4]
  Day 8 (2h) | 0.92 [0.5 to 1.3]
  Day 8 (4h) | 1.22 [0.7 to 2.2]
  Day 8 (6h) | 1.08 [0.8 to 1.7]
  Day 8 (8h) | 0.75 [0.6 to 1.1]
  Day 8 (12h) | 0.91 [0.6 to 1.5]
  Day 8 (24h) | 0.68 [0.4 to 1.0]

7. Secondary Outcome: Maximum Change From Baseline in Plasma Lactate Levels
Description: Lactate levels were analyzed in plasma samples collected during metformin alone or in combination with copanlisib. Maximum change from baseline on Day 1 and Day 8 was summarized.
Time Frame: From pre-dose up to 24 hours after study drug administration on Day 1 and Day 8
Population: Safety Analysis Set (SAF): included all participants who received at least one dose of the study medication.
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Copanlisib (Aliqopa, BAY80-6946) + Metformin
Number analyzed (Participants) | 13
mmol/L
  Day 1 (0.5h) | -0.04 [-0.4 to 0.3]
  Day 1 (1h) | 0.05 [-0.4 to 0.7]
  Day 1 (2h) | -0.04 [-0.4 to 0.3]
  Day 1 (4h) | 0.23 [-0.3 to 0.7]
  Day 1 (6h) | -0.03 [-0.5 to 0.5]
  Day 1 (8h) | 0.02 [-0.5 to 0.2]
  Day 1 (12h) | 0.26 [-0.1 to 1.6]
  Day 1 (24h) | 0.12 [-0.3 to 1.3]
  Day 8 (0h) | 0.01 [-0.4 to 0.2]
  Day 8 (0.5h) | 0.07 [-0.3 to 0.5]
  Day 8 (1h) | 0.12 [-0.3 to 0.6]
  Day 8 (2h) | 0.14 [-0.4 to 0.4]
  Day 8 (4h) | 0.44 [-0.3 to 1.2]
  Day 8 (6h) | 0.31 [-0.2 to 0.7]
  Day 8 (8h) | -0.02 [-0.4 to 0.1]
  Day 8 (12h) | 0.13 [-0.1 to 0.5]
  Day 8 (24h) | -0.10 [-0.5 to 0.1]

ADVERSE EVENTS:
Time Frame: From start of study medication until 30 days after end of treatment with study medication, up to 38 days.
Description: The study has only 1 arm with all subjects having received 2 doses on D1 (metformin alone) and D8 (metformin+ copanlisib).The study is not designed to compare the safety following 2 doses.
Arm/Group | Copanlisib (Aliqopa, BAY80-6946) + Metformin
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 11/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copanlisib (Aliqopa, BAY80-6946) + Metformin (N=13)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT03655301/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT03655301/SAP_001.pdf